CLINICAL TRIAL: NCT04829812
Title: Medical Compression for Leg Chronic Wound in Patients With Arterial Peripheral Disease: A Practice Survey
Brief Title: Medical Compression in Patients With Chronic Wound and Peripheral Arterial Disease
Acronym: COMPAD2
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Société Française de Médecine Vasculaire (SFMV) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0162
Record Dates: First submitted 2021-03-17; First posted 2021-04-02 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Peripheral Arterial Disease; Chronic Wound of the Lower Limb (Leg Ulcer or Foot Ulcer)
Keywords: compression system necessary; ankle brachial index; brachial index
MeSH Terms: conditions — Peripheral Arterial Disease; Leg Ulcer; Foot Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Prospective cohort with inclusion of consecutive or pseudo-consecutive patients by vascular specialist at their place of practice. Patient follow-up to assess wound progression and compression tolerance

SUMMARY:
Real-life practice survey of vascular specialist in France caring for patients with chronic wound for which compression treatment would be indicated and arterial disease of the lower limbs

DETAILED DESCRIPTION:
The leg chronic wound is a frequent and recurrent chronic disease of the lower limb, causing an impairment in the quality of life of patients and at a significant cost to society. Medical compression is essential for the healing of a leg ulcer.

However, the leg chronic wound is often associated with peripheral arterial disease (PAD), the prevalence of which in this population varies depending on the detection method used and the stage of arterial disease. The association of a chronic wound of the lower limb with PAD can occur two problems: the indication for compression and the validity of vascular explorations to detect arterial involvement and assess its severity.

The first issue concerns the use of compression in the presence of an PAD, which is the subject of controversy. Indeed, compression can improve tissue perfusion by reducing edema, but it carries a potential risk of ischemia and worsening of the ulcer, which probably increases with the progressive stage of PAD. Thus, medical compression is sometimes contraindicated, but the PAD severity threshold setting the contraindication varies from one recommendation to another.

The second problem concerns the validity of the detection and quantification methods of the PAD. Arterial involvement is probably underestimated by the clinic alone, in these patients whose mobility is sometimes reduced or who have trophic disorders of mixed origin, and the use of additional examinations (Doppler ultrasound, ankle or toe systolic pressures, TcPO2 or other vascular explorations) is necessary. There is no specific studies in the context of chronic wound of the lower limb (leg ulcer and foot ulcer) nevertheless hemodynamic measurements remain important to guide the indication (and the contraindication) for compression and the choice of the type of compression, suitable for each patient.

It seems important to evaluate this management charge by a practice investigation, in real life. Thus, the aim of this study is an observation of the real-life survey type of vasculars specialists in France caring for patients with a chronic wound of the lower limb (leg ulcer and foot ulcer) for which compression treatment would be indicated and arterial disease of the lower limbs. This is a prospective cohort with inclusion of consecutive or pseudo-consecutive patients by vascular specialist. Patients will be followed to ulcer development and tolerance of compression during 6 months.

ELIGIBILITY:
Inclusion criteria:

* Patient taken care of by a vascular specialist

  * Practicing, in a hospital or not or in a healing center,
  * Caring for patients with leg ulcers requiring the indication of compression treatment,
  * Can include consecutive patients at each consultation over the entire duration of the study or at a pre-established rate of at least half a day per week
* Patient with a chronic leg wound (leg ulcer and foot ulcer), defined as a chronic leg wound that does not spontaneously tend to heal after 6 weeks in the case of a first episode or 2 weeks in the case of recurrenceo In principle justifying a compression treatment, o And concomitantly presenting with PAD, retained by the investigator according to clinical and hemodynamic criteria that he will describe.

Exclusion criteria:

* Patient not giving his consent for collection of study data
* Patient with a life expectancy of less than 6 months.
* Patients for whom telephone follow-up is impossible (no contact possible with the patient, family and friends, IDE and the doctor)
* Patient presenting:
* A leg wound that is not chronic, or does not validate the ulcer criteria;
* An ulcer not located on the leg, in particular trophic disorders above the knee;
* Necrotic angiodermatitis
* Systemic sclerosis
* An infected ulcer (not temporary)
* An arterial ulcer, with PAD at the critical ischemia stage (ICC 2020 consensus), ABI<0.6, systolic ankle pression <60mmHg, systolic toe pression<30mmHg, TCPO2<20mmHg, bypass of lower limbs
* Patients for whom compression is not an option, regardless of arteriopathy, especially in cases of:

  * Allergy or intolerance to compression equipment
  * Practical or organizational installation difficulties
  * Morphotype difficult to fit (due to obesity, cachexia, trauma, dermatosis or other ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting: - a leg ulcer: these are incidental cases of leg ulcers with or without edema but giving rise to the benefit of compressive treatment. . Foot ulcer is not included. - PAD, the diagnosis of which is retained by the investigator, based on clinical and hemodynamic criteria, the method (s) and results of which he will specify.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Description of the practice of vascular specialist in the management of leg ulcers requiring medical compression | 1 day (inclusion visit)
  1. Description of the practice of vascular specialist in the management of chronic wound of lower limbs (CWOLL) requiring medical compression Methods do they use to detect and assess the severity of PAD: ( for example: ABI, TBI, USDuplex, pole test etc…) before the choice of de compression

SECONDARY OUTCOMES:
Efficacy and tolerance of this treatment | 6 months
  To prepare for future studies, markers of efficacy and tolerance of this treatment will be collected such as reduction of oedema (ankle circumference) , healing ulcer (planimetry), additional treatment (surgery, medical) and occurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Monira NOU, PHD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC